CLINICAL TRIAL: NCT07194330
Title: External Iliac Artery Endofibrosis: Performance-Related Suspicion, Diagnosis, Treatment, and Management in a Cyclist
Brief Title: External Iliac Artery Endofibrosis in Cycling
Status: Active, not recruiting | Type: Observational
Sponsor: Jesus Torres (Other)
Responsible Party: Sponsor-Investigator, Jesus Torres, Jesús Torres-Pérez: BsC, MD., University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Other Study IDs: M10/2025/304
Record Dates: First submitted 2025-08-05; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Iliac Artery Occlusive Disease; Blood Flow Velocity; Performance; Cycling
Keywords: External Iliac Artery; Endofibrosis; Cycling; Angiology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant with Iliac external endofibrosis disease: Participant will be recruited and information about his training and test in diagnosis process will be analysed.
  Interventions: Diagnostic Test: None-placebo

INTERVENTIONS:
Diagnostic Test: None-placebo — Not be displayed, only retrospective data will be required

SUMMARY:
A data request will be made regarding the tests conducted by the subject related to their performance, as well as the results of the medical diagnostic tests performed. The requested data/variables pertain to physical performance: power output on the pedals during training sessions, tests, and competitions, as well as medical tests during the diagnostic process.

DETAILED DESCRIPTION:
The medical tests include those performed during the diagnostic process of the pathophysiology of external iliac artery endofibrosis: imaging tests (Doppler ultrasound), exercise stress tests, computed tomography (CT) imaging, and intravascular ultrasound (IVUS). Data collection will be carried out prior to analysis and processing of the results; all data will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of external iliac artery endofibrosis confirmed by medical imaging (e.g., Doppler ultrasound, CT scan, or IVUS).

Age between 18 and 65 years.

Must be a regular cyclist (at least 500 training sessions per year for the past 5 years).

Ability to complete physical performance tests (e.g., cycling power output measurements, Lactate Threshold test).

No prior surgical intervention for external iliac artery endofibrosis or other lower extremity diseases

Willingness to provide informed consent and participate in the study.

Exclusion Criteria:

History of major cardiovascular disease (e.g., heart attack, stroke).

Pregnancy or breastfeeding.

Use of medications that significantly affect vascular health (e.g., anticoagulants, steroids).

Uncontrolled diabetes or other chronic metabolic disorders.

Recent lower extremity surgery (within the last 6 months).

Any condition that could interfere with the performance tests (e.g., neurological disorders, severe joint pain).

Diagnosis of other vascular diseases (e.g., deep vein thrombosis, atherosclerosis) that could affect arterial function.

History of systemic or local infections that may impact the vascular system.

History of significant trauma or injury to the lower extremities (e.g., fractures, ligament tears).

Any condition preventing safe participation in physical tests, including severe cardiovascular or musculoskeletal limitations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with the presence of external iliac artery endofibrosis pathophysiology, detected through performance-related suspicion, diagnosed, undergoing treatment, and in recovery
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Eco-Doppler with colour | 12 months pre-intervention/procedure/surgery; 12 months post-intervention/procedure/surgery.
  The results of distal systolic flow at rest and after a performance claudication test will be assessed. These will be measured using imaging to provide qualitative control of the results, as well as by evaluating the peak systolic flow velocity in the external iliac artery in centimeters per second (cm/s).
Performance data in training and competition | 3 years "pre" and 2 years "post intervention/surgery", and during study completion, a total of 5 years of time frame
  Data of power applied on pedals´powermeter will be collected, data will be from 2022 to 2025 training and competitive seasons, it will be collected as power in watts applied by cyclist during pedal stroke, conidered as external load.
  External load developed by participant during trainings and competitions will be collected in raw format, as watts applied by participant meassured by his powermeter installed in his bicycle second by second.
Distal systolic and dyastolic pressure | 12 months pre-intervention/procedure/surgery; 12 months post-intervention/procedure/surgery.
  Distal systolic and diastolic pressure will be assessed before and after a specific claudication test, and it will be recorded in millimeters of mercury (mmHg).
Angiography | 12 months pre-intervention/procedure/surgery
  The angiography test will be carried out using computed tomography and intravascular ultrasound examinations via catheterization. Imaging results from angiography will be collected, the thickness of the arterial wall will be measured in millimeters, and a qualitative structural assessment of the imaging will be performed."
Outcomes during surgery | Perioperative/Periprocedural
  During the surgery, the results obtained from the procedure, as well as the applied technique, will be presented, potentially in the form of images or explanatory diagrams of the process.
Lactate thresholds test | Through study completion, an average of 2 years".
  The lactate threshold test will be performed to assess the power (watts) developed by the participant. Data collected during this test will be analyzed alongside other study variables to understand the relationships between performance metrics and the diagnosis of the condition described.

CONTACTS AND LOCATIONS:
Locations (1):
- C San Bartolome 4, Estella-Lizarra, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon request and following approval by the ethics committee, and will be released in an anonymized form

REFERENCES:
- [Background] Mansour A, Murney S, Jordan K, Laperna L. Endofibrosis: an unusual cause of leg pain in an athlete. J Sports Med Phys Fitness. 2016 Jan-Feb;56(1-2):157-61. Epub 2015 Jul 3. PMID 26140352